CLINICAL TRIAL: NCT05219240
Title: Evaluation of Body Composition Improvement With Visceral Adiposity-Focused Anti-Obesity Telehealth Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: 20Lighter (Industry)
Responsible Party: Principal Investigator, Jessica W. Barnes, PhD, Principal Investigator, 20Lighter
Other Study IDs: 20L02
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Obesity; Cardiovascular Diseases; Metabolic Syndrome; Metabolic Disease
Keywords: visceral adiposity; BMI; body composition; obesity; cardiovascular disease; metabolic syndrome; metabolic disease
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Metabolic Syndrome; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Program participants
  Interventions: Other: 20Lighter Program

INTERVENTIONS:
Other: 20Lighter Program — Visceral Adiposity-Focused Anti-Obesity Telehealth Program

SUMMARY:
A retrospective review of body composition changes in patients who participate in a 9-week non-invasive intensive health care provider supervised weight loss program as an overall cohort and in sub-cohorts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age and older, who enroll in the weight loss program are eligible for inclusion of the data review.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Current treatment of cancer
* Major organ transplant with immunosuppressant medication,
* Adult with a strict vegetarian diet,
* Certain psychiatric conditions (schizophrenia, bipolar disorder, manic depression)
* Adults with a BMI < 25.0 and no cardiovascular or metabolic comorbidities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20Lighter program participants
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Bodyweight Change | Baseline to 90 days
  Change in bodyweight
Body Mass Index (BMI) Change | Baseline to 90 days
  Change in Body Mass Index (BMI)
Visceral Adiposity Change | Baseline to 90 days
  Change in Visceral Adiposity
Body Fat % Change | Baseline to 90 days
  Change in Body Fat %
Lean Body Mass Change | Baseline to 90 days
  Change in Lean Body Mass
Intracellular Fluid % Change | Baseline to 90 days
  Change in Intracellular Fluid %

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Barnes, PhD, Principal Investigator — 20Lighter
Locations (2):
- United States (2):
  - 20Lighter Telehealth Program, Little Rock, Arkansas
  - 20Lighter Telehealth Program, Cheyenne, Wyoming

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fryar CD, Carroll MD, Afful J. Prevalence of overweight, obesity, and severe obesity among children and adolescents aged 2-19 years: United States, 1963-1965 through 2017-2018. NCHS Health E-Stats. 2020.
- [Background] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Background] Anderson JW, Konz EC, Frederich RC, Wood CL. Long-term weight-loss maintenance: a meta-analysis of US studies. Am J Clin Nutr. 2001 Nov;74(5):579-84. doi: 10.1093/ajcn/74.5.579. PMID 11684524
- [Background] Balasubramanian P, Longo VD. Growth factors, aging and age-related diseases. Growth Horm IGF Res. 2016 Jun;28:66-8. doi: 10.1016/j.ghir.2016.01.001. Epub 2016 Jan 7. PMID 26883276
- [Background] Barnosky AR, Hoddy KK, Unterman TG, Varady KA. Intermittent fasting vs daily calorie restriction for type 2 diabetes prevention: a review of human findings. Transl Res. 2014 Oct;164(4):302-11. doi: 10.1016/j.trsl.2014.05.013. Epub 2014 Jun 12. PMID 24993615
- [Background] Bhutani S, Klempel MC, Kroeger CM, Trepanowski JF, Varady KA. Alternate day fasting and endurance exercise combine to reduce body weight and favorably alter plasma lipids in obese humans. Obesity (Silver Spring). 2013 Jul;21(7):1370-9. doi: 10.1002/oby.20353. Epub 2013 May 29. PMID 23408502
- [Background] Choi IY, Piccio L, Childress P, Bollman B, Ghosh A, Brandhorst S, Suarez J, Michalsen A, Cross AH, Morgan TE, Wei M, Paul F, Bock M, Longo VD. A Diet Mimicking Fasting Promotes Regeneration and Reduces Autoimmunity and Multiple Sclerosis Symptoms. Cell Rep. 2016 Jun 7;15(10):2136-2146. doi: 10.1016/j.celrep.2016.05.009. Epub 2016 May 26. PMID 27239035
- [Background] Collier R. Intermittent fasting: the science of going without. CMAJ. 2013 Jun 11;185(9):E363-4. doi: 10.1503/cmaj.109-4451. Epub 2013 Apr 8. No abstract available. PMID 23569168
- [Background] Di Biase S, Lee C, Brandhorst S, Manes B, Buono R, Cheng CW, Cacciottolo M, Martin-Montalvo A, de Cabo R, Wei M, Morgan TE, Longo VD. Fasting-Mimicking Diet Reduces HO-1 to Promote T Cell-Mediated Tumor Cytotoxicity. Cancer Cell. 2016 Jul 11;30(1):136-146. doi: 10.1016/j.ccell.2016.06.005. PMID 27411588
- [Background] Dorff TB, Groshen S, Garcia A, Shah M, Tsao-Wei D, Pham H, Cheng CW, Brandhorst S, Cohen P, Wei M, Longo V, Quinn DI. Safety and feasibility of fasting in combination with platinum-based chemotherapy. BMC Cancer. 2016 Jun 10;16:360. doi: 10.1186/s12885-016-2370-6. PMID 27282289
- [Background] Eshghinia S, Mohammadzadeh F. The effects of modified alternate-day fasting diet on weight loss and CAD risk factors in overweight and obese women. J Diabetes Metab Disord. 2013 Jan 9;12(1):4. doi: 10.1186/2251-6581-12-4. PMID 23497604
- [Background] Hoddy KK, Kroeger CM, Trepanowski JF, Barnosky A, Bhutani S, Varady KA. Meal timing during alternate day fasting: Impact on body weight and cardiovascular disease risk in obese adults. Obesity (Silver Spring). 2014 Dec;22(12):2524-31. doi: 10.1002/oby.20909. Epub 2014 Sep 24. PMID 25251676
- [Background] Horne BD, Muhlestein JB, Anderson JL. Health effects of intermittent fasting: hormesis or harm? A systematic review. Am J Clin Nutr. 2015 Aug;102(2):464-70. doi: 10.3945/ajcn.115.109553. Epub 2015 Jul 1. PMID 26135345
- [Background] Johnstone A. Fasting for weight loss: an effective strategy or latest dieting trend? Int J Obes (Lond). 2015 May;39(5):727-33. doi: 10.1038/ijo.2014.214. Epub 2014 Dec 26. PMID 25540982
- [Background] Klempel MC, Kroeger CM, Varady KA. Alternate day fasting (ADF) with a high-fat diet produces similar weight loss and cardio-protection as ADF with a low-fat diet. Metabolism. 2013 Jan;62(1):137-43. doi: 10.1016/j.metabol.2012.07.002. Epub 2012 Aug 11. PMID 22889512
- [Background] Longo VD, Panda S. Fasting, Circadian Rhythms, and Time-Restricted Feeding in Healthy Lifespan. Cell Metab. 2016 Jun 14;23(6):1048-1059. doi: 10.1016/j.cmet.2016.06.001. PMID 27304506
- [Background] Mattson MP, Allison DB, Fontana L, Harvie M, Longo VD, Malaisse WJ, Mosley M, Notterpek L, Ravussin E, Scheer FA, Seyfried TN, Varady KA, Panda S. Meal frequency and timing in health and disease. Proc Natl Acad Sci U S A. 2014 Nov 25;111(47):16647-53. doi: 10.1073/pnas.1413965111. Epub 2014 Nov 17. PMID 25404320
- [Background] Patterson RE, Laughlin GA, LaCroix AZ, Hartman SJ, Natarajan L, Senger CM, Martinez ME, Villasenor A, Sears DD, Marinac CR, Gallo LC. Intermittent Fasting and Human Metabolic Health. J Acad Nutr Diet. 2015 Aug;115(8):1203-12. doi: 10.1016/j.jand.2015.02.018. Epub 2015 Apr 6. No abstract available. PMID 25857868
- [Background] Varady KA, Bhutani S, Klempel MC, Kroeger CM, Trepanowski JF, Haus JM, Hoddy KK, Calvo Y. Alternate day fasting for weight loss in normal weight and overweight subjects: a randomized controlled trial. Nutr J. 2013 Nov 12;12(1):146. doi: 10.1186/1475-2891-12-146. PMID 24215592